CLINICAL TRIAL: NCT02364193
Title: Thoracic Fluid Assessment by Dynamic Contrast-enhanced Magnetic Resonance Imaging and Bioimpedance Spectroscopy: An Explorative Study in Healthy Subjects
Brief Title: Thoracic Fluid Assessment by Contrast-enhanced Magnetic Resonance Imaging and Bioimpedance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Ingeborg Herold, MD, Catharina Ziekenhuis Eindhoven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL50327.060.14
Record Dates: First submitted 2015-01-16; First posted 2015-02-18 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Congestion
Keywords: Intrathoracic blood volume; Extravascular lung water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thoracic fluid status assessment (Experimental): Cardiac MRI by a 1.5 Tesla scanner:
  * Left ventricular ejection fraction (LVEF), tracing short axis endocardial borders.
  * CO, phase contrast angiography.
  * Fluid challenge by auto-transfusion by distal leg compression using inflatable cuffs (Lympamat Digital Gradient system).
  * DCE-MRI, bolus injection of Gd-CA intravenously by an injector. Each subject will receive repeated injections (10% of maximum dose).
  * BIS, impedance will be measured continuously using ImpediMed-SFB7 and surface electrodes on the thorax. .
  Interventions: Device: MRI; Drug: Gd-CA; Device: BIS ImpediMed™ SFB7; Device: Autotransfusion Lympamat Digital Gradient system

INTERVENTIONS:
Device: MRI — Cardiac MRI for LVEF and segmentation.
  * Phase-contrast MRI for CO in aorta and each pulmonary vein.
  * DCE-MRI for bolus kinetic parameter analysis.
Drug: Gd-CA — Bolus kinetic parameter analysis, different doses of Gd-CA (Dotarem by Guerbet) ranging between 0.1 and 0.5 mmol will be injected intravenously after dilution in 5 milliliter saline by an injector at a speed of 5 ml/s.
Device: BIS ImpediMed™ SFB7 — BIS will be measured by Bio-impedance spectroscopy will be performed using ImpediMed™ SFB7 (ImpediMed Limited 2008).
  Impedance will be measured continuously during the fluid challenge and for maximum 600 seconds before and after the fluid challenge.
  Currents of different frequencies will be applied; the resulting voltage will be recorded, with a time resolution for the complete frequency span not lower than 2 seconds.
Device: Autotransfusion Lympamat Digital Gradient system — Lympamat Digital Gradient system (Bosl, Aachen) inflatable leg compression trousers will induce an autotransfusion by compressing the legs with a maximum of 90 mmHg for a maximum of 300 seconds

SUMMARY:
Heart failure (HF) is a major health problem, which is characterized by reduced cardiac function leading to pulmonary congestion. Most episodes of acute HF requiring unplanned hospitalization are due to pulmonary congestion. There is an urgent clinical need for quantitative, reproducible, minimally invasive, and noninvasive methods to assess thoracic fluid status. The potential value of dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) to this end has been suggested and demonstrated in-vitro. In this study the investigators aim to compare intra-thoracic fluid volume assessed by DCE- MRI using bolus kinetic parameters of the indicator dilution theory and bioimpedance spectroscopy (BIS).

Primary objectives: This study evaluates the correlation between change in BIS and change in bolus kinetic parameters in response to a fluid challenge.

Secondary objectives: The sensitivity of the bolus kinetic parameters to fluid challenges and the normal range DCE-MRI bolus kinetic parameters is evaluated in healthy subjects.

Study design: Prospective nonrandomized pilot study.

Study population: Healthy volunteers.

Intervention: The subjects will receive an intra-venous injection of gadolinium, a MRI contrast agent. External pressure will be applied by means of a leg-compression device in order to induce a rapid increase of the preload by blood auto-transfusion.

Main study parameters: Pulmonary transit time (PTT), skewness of the indicator dilution curve which is a measure of trans-pulmonary dilution, intrathoracic blood volume (ITBV), changes in bolus kinetic parameters, and thoracic impedance in response to fluid challenges. The correlation between changes in bolus kinetic parameters and thoracic impedance in response to fluid challenges.

DETAILED DESCRIPTION:
HF is a major health problem that affects 6.5 million people in Europe and 200.000 in the Netherlands. HF is characterized by frequent and often costly hospitalizations. Most hospitalizations for acute heart failure are due to pulmonary congestion rather than low cardiac output syndrome. Congestion is one of the clinical targets for current therapeutic approaches. Therefore, the assessment of fluid status is crucial for diagnosis, management, stratification and follow-up of HF patients.

Existing HF diagnostic tools:

Congestion is usually assessed by clinical signs such as dyspnea, oedema, rales, and jugular venous distension. Semi-quantitative scores have been developed, which may be used to follow-up response to HF therapy. However, these scores offer limited added clinical value because of the lack of an acceptable reproducibility, specificity, and sensitivity.

Indicator dilution theory and bolus kinetic analysis:

Assessment of congestion is possible by kinetic analysis of a bolus of a suitable indicator. Circulation tests based on this principle are well-known techniques to diagnose cardiac failure. Lower cardiac output (CO) and large lung blood volumes result in prolongation of circulation times.

Using the indicator dilution theory, bolus kinetic analysis can provide absolute volume measurement. The volume between injection and detection site or between different detection sites can be obtained by multiplying the difference in mean transit time of the indicator between the two sites and the flow rate of the dilution system. Furthermore, in case the indicator leaks from a membrane during the dilution process, kinetic parameters such as skewness of the indicator dilution curve may indicate the status of the membrane. The method was in principle applied by radionuclide angiography. Main limitations were the burden for the patient due to the use of radioactive tracers and the limitation of the method to the vessels, as it was not applicable for a large blood pool such as the heart ventricles. Other indicators such as dyes or cold saline require central vessel catheterization, an invasive procedure that results in severe additional risks for the patient.

DCE-MRI allows minimally invasive measurement of indicator dilution curves, with the advantage of simultaneous sampling in the different heart chambers. DCE-MRI has been proposed and validated in-vitro for volume measurement. It is a minimally invasive procedure that may advantage from automated post-processing techniques.

A small dose of gadolinium (Gd-CA) is used to ensure the linearity between the obtained MRI signal and the concentration of Gd-CA, for the indicator dilution theory. This bolus is much smaller than normally used for standard MRI protocols, this minimizes the risk for Gd-CA associated complications.

Compared to similar approaches in magnetic resonance angiography, DCE-MRI provides single heart beat resolution. Short post-processing time is required to derive physiological parameters since automated image processing and fitting routines are available.

Most studies focus only on left ventricle (LV) enhancement curve. This neglects right ventricle (RV) enhancement curve dilution system and therefore the hemodynamic status of the injection site to RV circulatory tree. Most studies only focus on the interpeak distance. A model-based curve fitting approach leads to more accurate results, not limited to the imaging sampling rate; which may lead to further estimation of additional parameters, possibly related to the lung circulation and its extravasation.

Pulmonary transit time (PTT) measured by DCE-MRI has been shown to be a good measure of preload and the LV filling pressure. The PTT was prolonged and correlated with alternative indirect congestion measures. Extravascular lung water (EVLW) currently can be assessed by chest X-ray, invasive thermodilution, or ultrasound comets. DCE-MRI based bolus kinetic offers a potential method for quantification of EVLW since due to their molecular weight, Gd-CAs are known to extravasate from the pulmonary circulation.

Impedance-based measurements:

An alternative approach to quantify thoracic fluids relies on transthoracic impedance measurements. These measurements can be performed non-invasive and continuous, which makes this a potential interesting monitoring tool for clinical practice to follow the trend of fluid redistribution towards pulmonary congestion. Previous evidences have shown that a decrease in thoracic impedance anticipates the need for hospitalization in HF patients.

Bio-impedance spectroscopy (BIS) is multi-frequency spectroscopy impedance measurement technique. All impedance-based measurements are limited to changes in volume and therefore need individual calibration to produce accurate absolute volumes. Moreover, several patient related characteristics, such as adiposity, height, and lung characteristics can also alter impedance-derived parameters. Therefore, because of the resultant high inter and intra-subject variability, only relative changes over time are significant. Impedance has been shown to be sensitive to fluid displacement in response to postural manoeuvres.

DCE-MRI and BIS provide complementary information. A monitoring strategy based on MRI at baseline and consecutive follow-up with BIS would satisfy the requirements for a clinically useful measurement technique that allows to reliably monitor the transition towards cardiopulmonary congestion even before clinical signs are present.

Goal of the study:

In this study the investigators aim to investigate whether changes in intrathoracic volumes can reliably be quantified by DCE-MRI and BIS measurements. The investigators hypothesize that such change in thoracic fluid distribution induced by fluid challenges can be detected in a minimally invasive way by DCE-MRI and by BIS, with agreement between the results of the two measurement techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Informed consent.
* Body mass index between 18 and 25

Exclusion Criteria:

* End-stage renal or hepatic disease
* Pregnancy
* Mild or moderate renal insufficiency, (GFR<60 mL/min);
* Risk for developing nephrogenic systemic fibrosis;
* General contra-indications to magnetic resonance imaging
* Pro-inflammatory state, vascular endothelial dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Bolus kinetic parameters using Contrast-enhanced-MRI and BIS | 30 minutes
  Correlation between changes in PTT and skewness of transpulmonary dilution system by DCE-MRI and changes in extravascular resistance measured by bio-impedance spectroscopy

SECONDARY OUTCOMES:
Fluid challenge response | 15 minutes
  Changes in PTT and skewness of transpulmonary dilution curve measured by DCE-MRI in response to fluid challenge/autotransfusion
Bolus kinetic parameters (Optimal DCE-MRI imaging sequence and range of normal values for ITBV, PTT and skewness of transpulmonary circulation measured by DCE-MRI in healthy subjects) | 5 minutes
  Optimal DCE-MRI imaging sequence and range of normal values for ITBV, PTT and skewness of transpulmonary circulation measured by DCE-MRI in healthy subjects.
Bolus kinetic parameters and hemodynamic parameters. | 5 minutes
  Correlation between ITBV, PTT and CMR functional parameters in volunteers by pearson correlation/linear regression- and Bland-Altman analyses. ITBV [milliliter] and PTT [seconds] will be correlated to the cardiac output [l/min], ejection fraction [%], and end-diastolic volume [ml] measured all by CMR.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Mischi, Msc PhD, Study Director — Eindhoven University of Technology
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, Netherlands